CLINICAL TRIAL: NCT01305213
Title: A Randomized Phase II Evaluation of Single-Agent Bevacizumab (NSC #704865) and Combination Bevacizumab With Fosbretabulin Tromethamine (CA4P) (NSC #752293) in the Treatment of Recurrent or Persistent Epithelial Ovarian, Fallopian Tube or Primary Peritoneal Carcinoma
Brief Title: Bevacizumab With or Without Fosbretabulin Tromethamine in Treating Patients With Recurrent or Persistent Ovarian Epithelial, Fallopian Tube, or Peritoneal Cavity Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02666; NCI-2011-02666 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000696220; GOG-0186I (Other: NRG Oncology); GOG-0186I (Other: CTEP); U10CA180868 (NIH); U10CA027469 (NIH)
Record Dates: First submitted 2011-02-25; First posted 2011-02-28 (Estimated); Results first posted 2017-07-12 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Recurrent Fallopian Tube Carcinoma; Recurrent Ovarian Carcinoma; Recurrent Primary Peritoneal Carcinoma
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — Bevacizumab; Immunoglobulin G; Disulfides

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (bevacizumab) (Active Comparator): Patients receive bevacizumab IV over 30-90 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Bevacizumab; Other: Laboratory Biomarker Analysis
- Arm II (bevacizumab, fosbretabulin tromethamine) (Experimental): Patients receive bevacizumab IV over 30-90 minutes and fosbretabulin tromethamine IV over 10-20 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Bevacizumab; Drug: Fosbretabulin Tromethamine; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Biological: Bevacizumab — Given IV
  Other Names: Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF rhuMAb; Avastin; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar CBT 124; Bevacizumab Biosimilar FKB238; Bevacizumab Biosimilar HD204; Bevacizumab Biosimilar HLX04; Bevacizumab Biosimilar IBI305; Bevacizumab Biosimilar LY01008; Bevacizumab Biosimilar MIL60; Bevacizumab Biosimilar QL 1101; Bevacizumab Biosimilar SCT501; HD204; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF; SCT501
Drug: Fosbretabulin Tromethamine — Given IV
  Other Names: CA4P; Zybrestat
  Arms: Arm II (bevacizumab, fosbretabulin tromethamine)
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This randomized phase II trial studies how well bevacizumab with or without fosbretabulin tromethamine works in treating patients with ovarian epithelial, fallopian tube, or peritoneal cavity cancer that has come back or is persistent. Monoclonal antibodies, such as bevacizumab, find tumor cells and help kill them. Bevacizumab and fosbretabulin tromethamine may stop the growth of ovarian cancer by blocking blood flow to the tumor. It is not yet known whether bevacizumab is more effective with or without fosbretabulin tromethamine in treating ovarian epithelial, fallopian tube, and peritoneal cavity cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the progression-free survival hazard ratio of the combination of bevacizumab and fosbretabulin tromethamine (CA4P) compared to bevacizumab alone in patients with persistent or recurrent ovarian, fallopian tube, or primary peritoneal cancer.

SECONDARY OBJECTIVES:

I. To determine the nature and degree of toxicity of fosbretabulin tromethamine plus bevacizumab.

II. To characterize and compare progression-free survival in patients with measurable disease (Response Evaluation Criteria in Solid Tumors [RECIST] criteria) and patients with detectable (non-measurable) disease between regimens.

III. To determine the overall survival for both regimens. IV. To estimate the proportion of patients with measurable disease who have objective tumor responses by treatment.

V. To provide descriptive information about cancer antigen (CA)-125 responses by regimen and where possible by objective tumor responses.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive bevacizumab intravenously (IV) over 30-90 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive bevacizumab IV over 30-90 minutes and fosbretabulin tromethamine IV over 10-20 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have recurrent or persistent epithelial ovarian, fallopian tube, or primary peritoneal carcinoma; histologic documentation of the original primary tumor is required via the pathology report
* Patients must have measurable disease or detectable (non-measurable) disease:

  * Measurable disease defined as at least one lesion that can be accurately measured in at least one dimension (longest dimension to be recorded); each lesion must be >= 10 mm when measured by computed tomography (CT) scan, magnetic resonance imaging (MRI) or caliper measurement by clinical exam, or >= 20 mm when measured by chest x-ray; lymph nodes must be >= 15 mm in short axis when measured by CT or MRI
  * Detectable disease in a patient is defined as one who does not have measurable disease but has at least one of the following conditions:

    * Baseline values of CA-125 at least 2 x upper limit of normal (ULN)
    * Ascites and/or pleural effusion attributed to tumor
    * Solid and/or cystic abnormalities on radiographic imaging that do not meet RECIST 1.1 definition for target lesions
* Patients in the measurable disease cohort must have at least one ?target lesion? to be used to assess response on this protocol as defined by RECIST 1.1; tumors within a previously irradiated field will be designated as ?non-target? lesions unless progression is documented or a biopsy is obtained to confirm persistence at least 90 days following completion of radiation therapy
* Patients must not be eligible for a higher priority Gynecologic Oncology Group (GOG) protocol, if one exists; in general, this would refer to any active GOG phase 3 protocol or rare tumor protocol for the same patient population
* Patients who have had one prior treatment must have a performance status of 0, 1, or 2
* Patients who have had two or three prior treatments must have a performance status of 0 or 1
* Patients should be free of acute hepatitis and active infection requiring parenteral antibiotics (with the exception of uncomplicated urinary tract infection [UTI])
* Recovery from the effects of recent surgery, radiotherapy, or chemotherapy

  * Any hormonal therapy directed at the malignant tumor must be discontinued at least one week prior to registration
  * Any other prior therapy directed at the malignant tumor, including chemotherapy, biological/targeted and immunologic agents, must be discontinued at least 3 weeks prior to registration (including small molecules and murine monoclonal antibodies); chimeric or human or humanized monoclonal antibodies (including bevacizumab) or vascular endothelial growth factor (VEGF) receptor fusion protein (including VEGF Trap/aflibercept) must be discontinued for at least 12 weeks prior to registration; no investigational therapy within 30 days prior to the first date of study treatment
  * Any prior radiation therapy must be discontinued at least 4 weeks prior to registration
* Prior therapy:

  * Patients must have had one prior platinum-based chemotherapeutic regimen for management of primary disease containing carboplatin, cisplatin, or another organoplatinum compound; this initial treatment may have included intraperitoneal therapy, consolidation, non-cytotoxic (biologic/targeted agents, such as bevacizumab) or extended therapy administered after surgical or non-surgical assessment
  * Patients are allowed to receive, but are not required to receive, two additional cytotoxic regimens for management of recurrent or persistent disease, with no more than 1 non-platinum, non-taxane regimen
  * Patients are allowed to receive, but are not required to receive, non-cytotoxic (biologic/targeted agents, such as bevacizumab) therapy as part of their primary treatment regimen; patients must have NOT received any non-cytotoxic therapy (biologic/targeted agents) for management of recurrent or persistent disease (e.g., GOG protocol 170 series drugs or bevacizumab)
  * For the purposes of this study, poly (adenosine diphosphate [ADP]-ribose) polymerase (PARP) inhibitors will be considered ?cytotoxic?, and prior treatment with PARP inhibitors for primary or recurrent disease WILL be allowed (either alone or in combination with chemotherapy)
* Patients with both platinum-sensitive and platinum-resistant disease are eligible; patients with platinum-refractory disease are NOT eligible; platinum-refractory disease is defined as patients who have progression of disease during the preceding platinum treatment

  * Definitions:

    * Platinum-free interval (PFI) is the period of time from the date of last platinum therapy to the date of progression (recurrence by CA-125, CT, etc.; CT is preferred) of disease or initiation of subsequent therapy (whichever occurs first); non-platinum maintenance therapy (e.g., extending taxane treatment) is excluded as a ?subsequent therapy;? if the patient?s last regimen used platinum, and she has NOT progressed before enrolling onto this study, then her PFI will be calculated from the date of last platinum therapy to the date of registration onto this study
    * PFI for the most recent platinum therapy will need to be calculated before enrollment onto this study for stratification purposes (i.e. balanced randomization)
    * Patients who have a PFI =< 182 days (26 weeks) are defined as ?platinum resistant;? patients who have 182 < PFI =< 365 days are defined as ?GOG platinum sensitive;? finally, patients with PFI > 365 days are defined as ?platinum sensitive?
* ANC greater than or equal to 1,500/mcl
* Platelets greater than or equal to 100,000/mcl
* Hemoglobin greater than or equal to 9 g/dL
* Creatinine less than or equal to 1.5 x institutional upper limit of normal (ULN)
* Potassium within the normal reference range for the laboratory; correction with supplements is acceptable
* Magnesium within the normal reference range for the laboratory; correction with supplements is acceptable
* Calcium within the normal reference range for the laboratory; correction with supplements is acceptable
* Bilirubin less than or equal to 1.5 x ULN
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) =< less than or equal to 3 x ULN
* Alkaline phosphatase less than or equal to 2.5 x ULN
* Prothrombin time (PT) such that international normalized ratio (INR) is less than or equal to 1.5 x ULN (or an in-range INR, usually between 2 and 3, if a patient is on a stable dose of therapeutic warfarin) and a partial thromboplastin time (PTT) less than or equal to 1.5 x ULN
* Urine protein should be screened by urine analysis; if protein is 2+ or higher, a 24-hour urine protein should be obtained and the level must be < 1,000 mg (< 1.0 g/24 hrs) for patient enrollment
* Patients of childbearing potential must have a negative serum pregnancy test prior to the study entry and be practicing an effective form of contraception
* Patients must have signed an approved informed consent and authorization permitting the release of personal health information
* Patients must meet pre-entry requirements

Exclusion Criteria:

* Patients who have received prior fosbretabulin tromethamine or any other vascular disrupting agent (VDA)
* Patients with other invasive malignancies, with the exception of non-melanoma skin cancer and other specific malignancies as noted below, are excluded if there is any evidence of other malignancy being present within the last three years; patients are also excluded if their previous cancer treatment contraindicates this protocol therapy
* Patients who have received prior radiotherapy to any portion of the abdominal cavity or pelvis OTHER THAN for the treatment of ovarian, fallopian tube or primary peritoneal cancer within the last three years are excluded; prior radiation for localized cancer of the breast, head and neck, or skin is permitted, provided that it was completed more than three years prior to registration, and the patient remains free of recurrent or metastatic disease
* Patients who have received prior chemotherapy for any abdominal or pelvic tumor OTHER THAN for the treatment of ovarian, fallopian tube or primary peritoneal cancer within the last three years are excluded; patients may have received prior adjuvant chemotherapy for localized breast cancer, provided that it was completed more than three years prior to registration, and the patient remains free of recurrent or metastatic disease
* Patients with serious non-healing wound, ulcer, or bone fracture; this includes history of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess within 90 days prior to the first date of study treatment
* Patients with active bleeding or pathologic conditions that carry high risk of bleeding, such as known bleeding disorder, coagulopathy, or tumor involving major vessels
* Patients with history or evidence upon physical examination of central nervous system (CNS) disease, including primary brain tumor, seizures not controlled with standard medical therapy, any brain metastases, or history of cerebrovascular accident (CVA, stroke), transient ischemic attack (TIA) or subarachnoid hemorrhage within six months prior to the first date of treatment on this study
* Patients with clinically significant cardiovascular disease; this includes:

  * Uncontrolled hypertension, defined as systolic > 150 mm Hg or diastolic > 90 mm Hg despite antihypertensive medications
  * History of torsade de pointes, ventricular tachycardia or fibrillation, pathologic sinus bradycardia (< 60 beats per minute [bpm]), heart block (excluding 1st degree block being, PR interval prolongation only), congenital long QT syndrome, new ST segment elevation or depression, or new Q waves on electrocardiogram (ECG)
  * Patients with corrected QT interval (QTc) > 470 msec
  * Requirement for receiving any drug known to prolong the QTc interval, including anti-arrhythmic medications; stable regimen of antidepressants of the selective serotonin reuptake inhibitor (SSRI) class is allowed
  * Myocardial infarction or unstable angina within 6 months prior to registration
  * New York Heart Association (NYHA) class II or greater congestive heart failure
  * Serious cardiac arrhythmia requiring medication; this does not include asymptomatic, atrial fibrillation with controlled ventricular rate
  * Patients who have received prior treatment with an anthracycline (including doxorubicin and or pegylated liposomal doxorubicin [Doxil; PLD]) must have an echocardiogram assessment and are excluded if they have an ejection fraction < 50%
  * Common Terminology Criteria for Adverse Events (CTCAE) grade 2 or greater peripheral vascular disease (at least brief [< 24 hrs] episodes of ischemia managed non-surgically and without permanent deficit)
* Known hypersensitivity to any of the components of fosbretabulin tromethamine or bevacizumab
* Major surgery within 28 days prior to the first date of study treatment
* Anticipation of need for major surgical procedures during the course of the study
* Core biopsy within 7 days prior to the first date of study treatment
* Patients with clinical symptoms or signs of gastrointestinal obstruction and patients who require parenteral hydration and/or nutrition; patients with bowel involvement on CT scan
* Patients with medical history or conditions not otherwise previously specified which in the opinion of the investigator should exclude participation in this study; the investigator can consult the Study Chair or Study Co-Chairs for uncertainty in this regard
* Patients who are pregnant or nursing

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2011-03-21 (Actual); Primary Completion 2016-08-20 (Actual); Study Completion 2016-11-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bradley J Monk, Principal Investigator — NRG Oncology
Locations (51):
- United States (51):
  - Saint Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - John Muir Medical Center-Concord Campus, Concord, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - SCL Health Lutheran Medical Center, Wheat Ridge, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Mercy Hospital, Miami, Florida
  - Northeast Georgia Medical Center-Gainesville, Gainesville, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Sudarshan K Sharma MD Limited-Gynecologic Oncology, Hinsdale, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Saint Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Maine Medical Center-Bramhall Campus, Portland, Maine
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - MedStar Franklin Square Medical Center/Weinberg Cancer Institute, Baltimore, Maryland
  - University of Massachusetts Memorial Health Care, Worcester, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Saint Dominic-Jackson Memorial Hospital, Jackson, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Washington University School of Medicine, St Louis, Missouri
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Summa Akron City Hospital/Cooper Cancer Center, Akron, Ohio
  - University of Cincinnati/Barrett Cancer Center, Cincinnati, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - Greenville Health System Cancer Institute-Eastside, Greenville, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin

REFERENCES:
- [Derived] Monk BJ, Sill MW, Walker JL, Darus CJ, Sutton G, Tewari KS, Martin LP, Schilder JM, Coleman RL, Balkissoon J, Aghajanian C. Randomized Phase II Evaluation of Bevacizumab Versus Bevacizumab Plus Fosbretabulin in Recurrent Ovarian, Tubal, or Peritoneal Carcinoma: An NRG Oncology/Gynecologic Oncology Group Study. J Clin Oncol. 2016 Jul 1;34(19):2279-86. doi: 10.1200/JCO.2015.65.8153. Epub 2016 May 23. PMID 27217446

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated on 3/21/2011 and closed on 4/22/2013
Groups:
- Arm I Bevacizumab: Bevacizumab 15mg/kg IV Day 1 every 3 weeks
- Arm II Bevacizumab + Fosbretabulin: Bevacizumab 15mg/kg IV Day 1 every 3 weeks plus fosbretabulin tromethamine 60mg/m2 IV Day 1 every 3 weeks
Period: Overall Study
Arm/Group | Arm I Bevacizumab | Arm II Bevacizumab + Fosbretabulin
Started | 53 | 54
Completed | 53 | 54
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I Bevacizumab | Arm II Bevacizumab + Fosbretabulin | Total
Number analyzed (Participants) | 53 | 54 | 107
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.3 (12) | 64.9 (10.3) | 64.6 (11.15)
Age, Customized [Count of Participants; unit: Participants]
  30 - 39 years | 2 | 0 | 2
  40 - 49 years | 3 | 5 | 8
  50 - 59 years | 12 | 12 | 24
  60 - 69 years | 19 | 15 | 34
  70 - 79 years | 13 | 19 | 32
  > = 80 years | 4 | 3 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 54 | 107
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: The time from randomization until disease progression, death, or date of last contact. Endpoints are progression or death. Patients who are not observed with an endpoint are censored.
Time Frame: For those patients whose disease can be evaluated by physical examination, progression was assessed prior to each 21 day cycle. CT scan or MRI if used to follow lesion for measurable disease every other cycle, up to 5 years
Population: All intent to treat patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I Bevacizumab | Arm II Bevacizumab + Fosbretabulin
Number analyzed (Participants) | 53 | 54
months | 4.83 [4.14 to 6.24] | 7.23 [4.30 to 10.51]

2. Secondary Outcome: Incidence of Adverse Events (Grade 3 or Higher) as Assessed by Common Terminology Criteria for Adverse Events (CTCAE) v 4.0
Description: Toxicities will be characterized by their frequency and severity. Differences in the level of toxicities by treatment regimen will be assessed by classifying them as severe or not severe and examining the relative proportion of severe toxicities.
Time Frame: Up to 5 years
Population: All eligible and treated patients
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I Bevacizumab | Arm II Bevacizumab + Fosbretabulin
Number analyzed (Participants) | 53 | 54
Participants
  Thrombocytopenia | 0 | 1
  Neutropenia | 3 | 1
  Other Investigations | 1 | 4
  Other Blood/Lymphatics | 0 | 1
  Cardiac | 1 | 1
  Nausea | 2 | 3
  Vomiting | 0 | 2
  Other Gastrointestinal | 5 | 8
  General and Administration Site | 2 | 3
  Infections/Infestations | 3 | 3
  Metabolism/Nutrition | 8 | 11
  Musculoskeletal/Connective tissue | 2 | 2
  Neoplasms Benign/Malignant | 1 | 0
  Peripheral sensory Neuropathy | 0 | 1
  Nervous system | 1 | 2
  Renal/Urinary | 0 | 2
  Respiratory/Thoracic/Mediastinal | 2 | 1
  Vascular Disorders | 10 | 19

3. Secondary Outcome: Measurable Disease by Response Evaluation Criteria in Solid Tumors (RECIST) Criteria and Progression Free Survival (PFS)
Description: Differences between measurable versus non-measurable disease status on PFS and OS will be examined with plots of survival curves, estimates of quartiles and hazard ratios.
Time Frame: Up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Non Measurable Disease Patients: Patients with non measurable disease
- Measurable Disease Patients: Patients with measurable disease
Arm/Group | Non Measurable Disease Patients | Measurable Disease Patients
Number analyzed (Participants) | 26 | 81
months | 3.99 [2.73 to 5.19] | 6.80 [5.29 to 8.67]

4. Secondary Outcome: Tumor Response
Description: Complete and Partial Tumor Response by RECIST 1.0
Time Frame: for those patients whose disease can be evaluated by physical examination, response wa assessed prior to each 21 day cycle. CT scan or MRI if used to follow lesion for measurable disease every other cycle, up to 5 years
Population: Patients with measurable disease
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I Bevacizumab | Arm II Bevacizumab + Fosbretabulin
Number analyzed (Participants) | 39 | 42
percentage of participants | 28.2 [16.7 to 42.3] | 35.7 [23.5 to 49.5]

5. Secondary Outcome: Overall Survival (OS)
Description: as for outcome 3
Time Frame: Up to 5 years
Measure: Median (90% Confidence Interval); unit: months
Groups:
- Non Measurble Disease: Patients with non measurable disease
Arm/Group | Non Measurble Disease | Measurable Disease Patients
Number analyzed (Participants) | 26 | 81
months | 22.0 [13.3 to NA] — The proportion of patients who died at the time of the analysis was insufficient to estimate the upper bound of the confidence interval. | 21.2 [19.8 to NA] — The proportion of patients who died at the time of the analysis was insufficient to estimate the upper bound of the confidence interval.

6. Secondary Outcome: Response by CA-125
Description: The effects of treatment on the proportion responding by CA125 will be examined.
Time Frame: Up to 5 years
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Arm I Bevacizumab | Arm II Bevacizumab + Fosbretabulin
Number analyzed (Participants) | 38 | 27
Percentage of Participants | 23.7 [11.4 to 40.2] | 33.3 [16.5 to 54.0]

ADVERSE EVENTS:
Time Frame: All adverse Events (AEs) occurring during treatment and up to 30 days after stopping the study treatment are reported. Also reported are Serious Adverse Events (SAEs) considered to be treatment related for up to 5 years after stopping study treatment.
Arm/Group | Arm I Bevacizumab | Arm II Bevacizumab + Fosbretabulin
Serious Adverse Events (participants affected / at risk) | 9/53 | 16/54
Other Adverse Events (participants affected / at risk) | 53/53 | 52/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I Bevacizumab (N=53) | Arm II Bevacizumab + Fosbretabulin (N=54)
Atrial Fibrillation (Cardiac disorders) | 0 | 2
Chest Pain - Cardiac (Cardiac disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 1
Obstruction Gastric (Gastrointestinal disorders) | 0 | 1
Gastrointestinal Disorders - Other (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 0
Gastrointestinal Fistula (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Pleural Infection (Infections and infestations) | 1 | 0
Pelvic Infection (Infections and infestations) | 0 | 1
Device Related Infection (Infections and infestations) | 0 | 1
Inr Increased (Investigations) | 1 | 0
Electrocardiogram Qt Corrected Interval Prolonged (Investigations) | 0 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Neoplasms Benign, Malignant And Unspecified (Incl (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1
Thromboembolic Event (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I Bevacizumab (N=53) | Arm II Bevacizumab + Fosbretabulin (N=54)
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 23 | 19
Atrial Fibrillation (Cardiac disorders) | 0 | 2
Sinus Bradycardia (Cardiac disorders) | 1 | 3
Palpitations (Cardiac disorders) | 5 | 4
Sinus Tachycardia (Cardiac disorders) | 0 | 2
Chest Pain - Cardiac (Cardiac disorders) | 1 | 1
Tinnitus (Ear and labyrinth disorders) | 5 | 3
Hearing Impaired (Ear and labyrinth disorders) | 5 | 3
Ear Pain (Ear and labyrinth disorders) | 3 | 2
Eye Disorders - Other (Eye disorders) | 1 | 0
Watering Eyes (Eye disorders) | 2 | 0
Flashing Lights (Eye disorders) | 2 | 1
Eye Pain (Eye disorders) | 1 | 0
Photophobia (Eye disorders) | 0 | 1
Blurred Vision (Eye disorders) | 4 | 7
Dry Eye (Eye disorders) | 0 | 1
Floaters (Eye disorders) | 3 | 2
Dysphagia (Gastrointestinal disorders) | 2 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 5
Dry Mouth (Gastrointestinal disorders) | 0 | 5
Colonic Obstruction (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 16 | 25
Diarrhea (Gastrointestinal disorders) | 16 | 21
Vomiting (Gastrointestinal disorders) | 8 | 17
Bloating (Gastrointestinal disorders) | 6 | 7
Stomach Pain (Gastrointestinal disorders) | 1 | 2
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 3
Abdominal Pain (Gastrointestinal disorders) | 19 | 22
Rectal Hemorrhage (Gastrointestinal disorders) | 1 | 4
Oral Dysesthesia (Gastrointestinal disorders) | 1 | 3
Mucositis Oral (Gastrointestinal disorders) | 7 | 10
Lower Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 0 | 1
Oral Pain (Gastrointestinal disorders) | 0 | 4
Abdominal Distension (Gastrointestinal disorders) | 3 | 3
Nausea (Gastrointestinal disorders) | 22 | 22
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 3 | 2
Rectal Pain (Gastrointestinal disorders) | 1 | 0
Esophageal Ulcer (Gastrointestinal disorders) | 0 | 1
Fecal Incontinence (Gastrointestinal disorders) | 1 | 1
Hemorrhoidal Hemorrhage (Gastrointestinal disorders) | 0 | 1
Hemorrhoids (Gastrointestinal disorders) | 0 | 1
Tooth Development Disorder (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 4 | 2
Toothache (Gastrointestinal disorders) | 0 | 2
Dental Caries (Gastrointestinal disorders) | 0 | 1
Flatulence (Gastrointestinal disorders) | 1 | 2
General Disorders And Administration Site Conditio (General disorders) | 1 | 0
Pain (General disorders) | 7 | 14
Malaise (General disorders) | 2 | 1
Localized Edema (General disorders) | 1 | 0
Flu Like Symptoms (General disorders) | 0 | 3
Non-Cardiac Chest Pain (General disorders) | 0 | 3
Edema Limbs (General disorders) | 9 | 0
Fatigue (General disorders) | 35 | 42
Fever (General disorders) | 4 | 8
Gait Disturbance (General disorders) | 0 | 2
Chills (General disorders) | 0 | 4
Infusion Related Reaction (General disorders) | 0 | 2
Allergic Reaction (Immune system disorders) | 0 | 1
Infections And Infestations - Other (Infections and infestations) | 1 | 2
Wound Infection (Infections and infestations) | 2 | 1
Upper Respiratory Infection (Infections and infestations) | 2 | 2
Tooth Infection (Infections and infestations) | 1 | 1
Skin Infection (Infections and infestations) | 2 | 1
Sinusitis (Infections and infestations) | 4 | 2
Rash Pustular (Infections and infestations) | 0 | 1
Papulopustular Rash (Infections and infestations) | 0 | 1
Mucosal Infection (Infections and infestations) | 0 | 1
Device Related Infection (Infections and infestations) | 1 | 0
Gum Infection (Infections and infestations) | 0 | 1
Vaginal Infection (Infections and infestations) | 1 | 1
Urinary Tract Infection (Infections and infestations) | 10 | 7
Bronchial Infection (Infections and infestations) | 2 | 2
Injury, Poisoning And Procedural Complications - O (Injury, poisoning and procedural complications) | 1 | 2
Fracture (Injury, poisoning and procedural complications) | 1 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Wound Complication (Injury, poisoning and procedural complications) | 1 | 1
Bruising (Injury, poisoning and procedural complications) | 4 | 1
Investigations - Other (Investigations) | 1 | 1
Weight Loss (Investigations) | 8 | 6
Weight Gain (Investigations) | 1 | 0
Platelet Count Decreased (Investigations) | 6 | 10
Lymphocyte Count Decreased (Investigations) | 4 | 2
Inr Increased (Investigations) | 0 | 2
Electrocardiogram Qt Corrected Interval Prolonged (Investigations) | 0 | 4
Creatinine Increased (Investigations) | 10 | 3
Cholesterol High (Investigations) | 1 | 0
Cardiac Troponin T Increased (Investigations) | 1 | 0
Neutrophil Count Decreased (Investigations) | 7 | 8
Cardiac Troponin I Increased (Investigations) | 0 | 1
Blood Bilirubin Increased (Investigations) | 2 | 4
White Blood Cell Decreased (Investigations) | 11 | 8
Aspartate Aminotransferase Increased (Investigations) | 8 | 11
Alkaline Phosphatase Increased (Investigations) | 4 | 8
Alanine Aminotransferase Increased (Investigations) | 3 | 6
Activated Partial Thromboplastin Time Prolonged (Investigations) | 0 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 2 | 2
Hyponatremia (Metabolism and nutrition disorders) | 12 | 9
Hypomagnesemia (Metabolism and nutrition disorders) | 15 | 13
Hypokalemia (Metabolism and nutrition disorders) | 8 | 6
Hypoglycemia (Metabolism and nutrition disorders) | 4 | 4
Hypocalcemia (Metabolism and nutrition disorders) | 8 | 10
Hypoalbuminemia (Metabolism and nutrition disorders) | 10 | 9
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 | 0
Hypernatremia (Metabolism and nutrition disorders) | 2 | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 2 | 6
Hyperkalemia (Metabolism and nutrition disorders) | 7 | 4
Hyperglycemia (Metabolism and nutrition disorders) | 17 | 16
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 3
Anorexia (Metabolism and nutrition disorders) | 9 | 13
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 9 | 9
Neck Pain (Musculoskeletal and connective tissue disorders) | 3 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 14
Muscle Weakness Upper Limb (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle Weakness Lower Limb (Musculoskeletal and connective tissue disorders) | 1 | 2
Joint Range Of Motion Decreased (Musculoskeletal and connective tissue disorders) | 1 | 0
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 3 | 5
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Buttock Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 12 | 5
Arthritis (Musculoskeletal and connective tissue disorders) | 4 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 23 | 17
Tumor Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Nervous System Disorders - Other (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 1 | 1
Peripheral Sensory Neuropathy (Nervous system disorders) | 26 | 24
Peripheral Motor Neuropathy (Nervous system disorders) | 2 | 2
Paresthesia (Nervous system disorders) | 0 | 1
Neuralgia (Nervous system disorders) | 1 | 1
Memory Impairment (Nervous system disorders) | 2 | 2
Movements Involuntary (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 18 | 21
Extrapyramidal Disorder (Nervous system disorders) | 0 | 1
Dysphasia (Nervous system disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 3 | 1
Syncope (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 4 | 6
Cognitive Disturbance (Nervous system disorders) | 0 | 2
Ataxia (Nervous system disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 5 | 11
Depression (Psychiatric disorders) | 8 | 10
Confusion (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 9 | 7
Urinary Urgency (Renal and urinary disorders) | 0 | 2
Urinary Retention (Renal and urinary disorders) | 1 | 2
Urinary Incontinence (Renal and urinary disorders) | 4 | 4
Urinary Tract Pain (Renal and urinary disorders) | 5 | 4
Urinary Frequency (Renal and urinary disorders) | 4 | 3
Proteinuria (Renal and urinary disorders) | 9 | 6
Hematuria (Renal and urinary disorders) | 2 | 0
Chronic Kidney Disease (Renal and urinary disorders) | 1 | 1
Acute Kidney Injury (Renal and urinary disorders) | 1 | 0
Vaginal Pain (Reproductive system and breast disorders) | 0 | 1
Vaginal Hemorrhage (Reproductive system and breast disorders) | 1 | 4
Pelvic Pain (Reproductive system and breast disorders) | 3 | 2
Vaginal Discharge (Reproductive system and breast disorders) | 0 | 1
Breast Pain (Reproductive system and breast disorders) | 0 | 1
Respiratory, Thoracic And Mediastinal Disorders - (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Voice Alteration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Sinus Disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Postnasal Drip (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 3 | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 11 | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 17 | 15
Cough (Respiratory, thoracic and mediastinal disorders) | 17 | 10
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchopulmonary Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 8 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 2
Rash Acneiform (Skin and subcutaneous tissue disorders) | 1 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 6
Palmar-Plantar Erythrodysesthesia Syndrome (Skin and subcutaneous tissue disorders) | 0 | 1
Pain Of Skin (Skin and subcutaneous tissue disorders) | 0 | 1
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 3 | 7
Nail Loss (Skin and subcutaneous tissue disorders) | 0 | 2
Nail Discoloration (Skin and subcutaneous tissue disorders) | 1 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 1
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 0 | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 2 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 5 | 9
Thromboembolic Event (Vascular disorders) | 0 | 1
Lymphedema (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 2 | 3
Hypertension (Vascular disorders) | 28 | 32
Hot Flashes (Vascular disorders) | 1 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less